CLINICAL TRIAL: NCT07400146
Title: Instillation of Bupivacaine With Epinephrine Over Diaphragm to Reduce Postoperative Shoulder Pain Following Benign Gynecologic Laparoscopic Surgery: A Randomized Control Trial
Brief Title: Bupivacaine With Epinephrine Over Diaphragm in Laparoscopy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kelly Wright, Division Director of Minimally Invasive Gynecologic Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003947
Record Dates: First submitted 2026-01-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain; Shoulder Pain
Keywords: Laparoscopy; Gynecologic surgery; Bupivacaine
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trial, single blind study
Who Masked: Participant
Masking Description: Participants are randomized into either the treatment arm with placement of bupivacaine with epinephrine over the diaphragm or the no intervention arm. Participants are blinded to whether or not they received the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine with epinephrine (Experimental): Participants randomized to this arm will have 30 mL of 0.25% bupivacaine with epinephrine 1:200,000 (total of 75 mg) placed over the diaphragm laparoscopically at the conclusion of the laparoscopic gynecologic procedure.
  Interventions: Drug: Instillation of Bupivacaine with epinephrine over the diaphragm
- No intervention (No Intervention): No additional intervention will be performed.

INTERVENTIONS:
Drug: Instillation of Bupivacaine with epinephrine over the diaphragm — Prior to desufflation of the abdomen during the laparoscopic gynecologic procedure, the surgeon will instill 30mL of 0.25% bupivacaine with epinephrine 1:200,000 (total of 75 mg) laparoscopically aiming to cover the diaphragm with liquid.
  Arms: Bupivacaine with epinephrine

SUMMARY:
Postoperative shoulder pain is often reported to be particularly bothersome after laparoscopy. The benefits of local anesthetic, such as bupivacaine, applied to subcutaneous tissue for general postoperative pain management after surgery is well established. However, there have been no studies on sprayed bupivacaine over the diaphragm to reduce shoulder pain in laparoscopic surgery. The purpose of the study is to evaluate if sprayed infra-diaphragmatic bupivacaine compared to placebo (saline) will improve postoperative shoulder pain in patients undergoing benign laparoscopic gynecologic surgery. The entire study will be conducted at Cedar Sinai Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 8 years of age or older
* Undergoing laparoscopic surgery at Cedars-Sinai Medical Center with a surgeon in the Minimally Invasive Gynecologic Surgery division.

Exclusion Criteria:

* Pregnancy
* Urgent/non-scheduled surgery
* Scheduled for planned or possible concomitant non-gynecologic surgery (e.g., urologic or colorectal procedure)
* Baseline shoulder pain
* Baseline opioid use
* Baseline of chronic pain syndrome
* Conversion to open surgery
* Allergy or intolerance to bupivacaine, lidocaine (or amide class of anesthetics), oxycodone, acetaminophen, or ibuprofen
* Planned post-operative admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative shoulder pain scores | 24 hours postoperatively
  Reported right shoulder pain score using visual analog score (VAS) 24 hours postoperatively Null hypothesis = pain scores will not differ among the bupivacaine with epinephrine vs no intervention group Alternative hypothesis = pain scores will be lower among the bupivacaine with epinephrine group
  Assessed using the validated 100-mm scale with a range of 0-10 (11-point numerical rating scale), an ordinal scale Analyzed using the Kruskall Wallis test (as the data from the scale is typically not normally distributed); pairwise analyses will then be conducted using the Dunn post-hoc test if statistically significant Assuming non-normality, data will be presented as median (range) Patients without any postoperative documentation of pain scores will be withdrawn from the study and thus excluded from the analysis

SECONDARY OUTCOMES:
Post-operative generalized pain scores | up to 6 hours in post-anaesthesia care unit (PACU)
  Post-operative generalized pain scores (superiority):
  Null hypothesis = pain scores will not differ among the bupivacaine with epinephrine vs no intervention group Alternative hypothesis= pain scores will be lower among the bupivacaine with epinephrine group
  First and last reported generalized pain score in post-anaesthesia care unit (PACU) using numerical rating score Assessed using the validated 11-point numerical rating scale (0-10), an ordinal scale Analyzed using the Kruskall Wallis test (as the data from the scale is typically not normally distributed); pairwise analyses will then be conducted using the Dunn post-hoc test if statistically significant Assuming non-normality, data will be presented as median (range) Patients without any postoperative documentation of pain scores will be withdrawn from the study and thus excluded from the analysis
Total analgesic requirements in post-anaesthesia care unit (PACU) in morphine equivalents | up to 6 hours in post-anaesthesia care unit (PACU)
  Calculated in morphine milligram equivalents (continuous data) Analyzed using the Kruskall-Wallis test (assuming non-normal data) Data will be presented as median (range)
Length of stay in post-anaesthesia care unit (PACU) | up to 6 hours in post-anaesthesia care unit (PACU)
  Length of stay in post-anaesthesia care unit (PACU) (superiority):
  Null hypothesis = PACU length of stay will not differ among the bupivacaine with epinephrine vs no intervention group Alternative hypothesis= PACU length of stay will be shorter in the bupivacaine with epinephrine groups
  Documented in minutes (continuous data) Analyzed using ANOVA if normally distributed, Kruskall-Wallis test if not normally distributed
Post-operative shoulder pain scores at home | 5 days postoperatively
  Daily reported post-operative shoulder pain scores at home (superiority):
  Null hypothesis = pain scores will not differ among the bupivacaine with epinephrine vs no intervention group Alternative hypothesis = pain scores will be lower among the bupivacaine with epinephrine group
  Assessed using the validated 100-mm scale with a range of 0-10 (11-point numerical rating scale), an ordinal scale Analyzed using the Kruskall Wallis test (as the data from the scale is typically not normally distributed); pairwise analyses will then be conducted using the Dunn post-hoc test if statistically significant Assuming non-normality, data will be presented as median (range) Patients without any postoperative documentation of pain scores will be withdrawn from the study and thus excluded from the analysis
Post-operative opioid use | 1 week postoperative
  Post-operative opioid use (superiority):
  Null hypothesis = post-op opioid use will not differ among the bupivacaine with epinephrine vs no intervention group Alternative hypothesis= post-op opioid use will be lower among the bupivacaine with epinephrine group
  Number of pills used reported by patient (interval data) Analyzed using the Kruskall-Wallis test Data will be presented as median (range)
Surgical outcome: EBL | up to 8 hours
  Surgical outcomes: EBL (mL) Null hypothesis = outcome will not differ between groups Alternative hypothesis = outcome will be improved in bupivacaine with epinephrine group
  Continuous variables: estimated blood loss Analyzed using ANOVA if normally distributed, Kruskall-Wallis test if not normally distributed
Surgical outcome: operative time | up to 8 hours
  Surgical outcomes: operative time (minutes) Null hypothesis = outcome will not differ between groups Alternative hypothesis = outcome will be improved in bupivacaine with epinephrine group
  Continuous variables: operative time, estimated blood loss Analyzed using ANOVA if normally distributed, Kruskall-Wallis test if not normally distributed
Surgical outcome: intraoperative complications | within 1 week of surgery
  Surgical outcomes: intraoperative complications Null hypothesis = outcome will not differ between groups Alternative hypothesis = outcome will be improved in bupivacaine with epinephrine group
  Binary data: Surgical complications (yes/no) Analyzed using chi-square test
Surgical outcomes: conversion to laparotomy | within 6 hours of surgery start time
  Surgical outcomes: conversion to laparotomy Null hypothesis = outcome will not differ between groups Alternative hypothesis = outcome will be improved in bupivacaine with epinephrine group
  Binary data: conversion to laparotomy (yes/no) Analyzed using chi-square test

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammer A, Rositch AF, Kahlert J, Gravitt PE, Blaakaer J, Sogaard M. Global epidemiology of hysterectomy: possible impact on gynecological cancer rates. Am J Obstet Gynecol. 2015 Jul;213(1):23-29. doi: 10.1016/j.ajog.2015.02.019. Epub 2015 Feb 25. PMID 25724402
- [Background] Alperin M, Kivnick S, Poon KY. Outpatient laparoscopic hysterectomy for large uteri. J Minim Invasive Gynecol. 2012 Nov-Dec;19(6):689-94. doi: 10.1016/j.jmig.2012.06.007. PMID 23084671
- [Background] Driessen SR, Baden NL, van Zwet EW, Twijnstra AR, Jansen FW. Trends in the implementation of advanced minimally invasive gynecologic surgical procedures in the Netherlands. J Minim Invasive Gynecol. 2015 May-Jun;22(4):642-7. doi: 10.1016/j.jmig.2015.01.026. Epub 2015 Feb 3. PMID 25655043
- [Background] Johnson N, Barlow D, Lethaby A, Tavender E, Curr E, Garry R. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD003677. doi: 10.1002/14651858.CD003677.pub3. PMID 16625589
- [Background] Jaschinski T, Mosch C, Eikermann M, Neugebauer EA. Laparoscopic versus open appendectomy in patients with suspected appendicitis: a systematic review of meta-analyses of randomised controlled trials. BMC Gastroenterol. 2015 Apr 15;15:48. doi: 10.1186/s12876-015-0277-3. PMID 25884671
- [Background] Lirk P, Thiry J, Bonnet MP, Joshi GP, Bonnet F; PROSPECT Working Group. Pain management after laparoscopic hysterectomy: systematic review of literature and PROSPECT recommendations. Reg Anesth Pain Med. 2019 Apr;44(4):425-436. doi: 10.1136/rapm-2018-100024. Epub 2019 Feb 3. PMID 30914471
- [Background] Vadivelu N, Mitra S, Narayan D. Recent advances in postoperative pain management. Yale J Biol Med. 2010 Mar;83(1):11-25. PMID 20351978
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Bougie O, Blom J, Zhou G, Murji A, Thurston J. Use and misuse of opioid after gynecologic surgery. Best Pract Res Clin Obstet Gynaecol. 2022 Dec;85(Pt B):23-34. doi: 10.1016/j.bpobgyn.2022.07.005. Epub 2022 Jul 18. PMID 35973919
- [Background] Blanton E, Lamvu G, Patanwala I, Barron KI, Witzeman K, Tu FF, As-Sanie S. Non-opioid pain management in benign minimally invasive hysterectomy: A systematic review. Am J Obstet Gynecol. 2017 Jun;216(6):557-567. doi: 10.1016/j.ajog.2016.12.175. Epub 2016 Dec 30. PMID 28043841
- [Background] Clark NV, Moore K, Maghsoudlou P, North A, Ajao MO, Einarsson JI, Louie M, Schiff L, Moawad G, Cohen SL, Carey ET. Superior Hypogastric Plexus Block to Reduce Pain After Laparoscopic Hysterectomy: A Randomized Controlled Trial. Obstet Gynecol. 2021 Apr 1;137(4):648-656. doi: 10.1097/AOG.0000000000004329. PMID 33706344
- [Background] Miao L, Chen Q, Wang Y, Wang D, Zhou M. Effect of intraperitoneal infusion of ropivacaine combined with dexmedetomidine in patients undergoing total laparoscopic hysterectomy: a single-center randomized double-blinded controlled trial. Arch Gynecol Obstet. 2024 Apr;309(4):1387-1393. doi: 10.1007/s00404-023-07020-w. Epub 2023 Apr 1. PMID 37004537
- [Background] Patel R, Carvalho JC, Downey K, Kanczuk M, Bernstein P, Siddiqui N. Intraperitoneal Instillation of Lidocaine Improves Postoperative Analgesia at Cesarean Delivery: A Randomized, Double-Blind, Placebo-Controlled Trial. Anesth Analg. 2017 Feb;124(2):554-559. doi: 10.1213/ANE.0000000000001799. PMID 27984226
- [Background] Cho M, Kim CJ, Hahm TS, Lee YY, Kim TJ, Lee JW, Kim BG, Bae DS, Choi CH. Combination of a pulmonary recruitment maneuver and intraperitoneal bupivacaine for the reduction of postoperative shoulder pain in gynecologic laparoscopy: a randomized, controlled trial. Obstet Gynecol Sci. 2020 Mar;63(2):187-194. doi: 10.5468/ogs.2020.63.2.187. Epub 2020 Feb 20. PMID 32206659
- [Background] Sutchritpongsa P, Chaipakdi P, Sirimai K, Chalermchokcharoenkit A, Tanmahasamut P. Intraperitoneal sub-diaphragmatic instillation of bupivacaine plus morphine for reducing postoperative shoulder pain after gynecologic endoscopy. J Med Assoc Thai. 2013 May;96(5):513-8. PMID 23745303
- [Background] Roy KK, Subbaiah M, Naha M, Kumar S, Sharma JB, Jahagirdar N. Intraperitoneal bupivacaine for pain relief after minilaparoscopy in patients with infertility. Arch Gynecol Obstet. 2014 Feb;289(2):337-40. doi: 10.1007/s00404-013-2994-6. Epub 2013 Aug 8. PMID 23925646
- [Background] Ruiz-Tovar J, Gonzalez J, Garcia A, Cruz C, Rivas S, Jimenez M, Ferrigni C, Duran M. Intraperitoneal Ropivacaine Irrigation in Patients Undergoing Bariatric Surgery: a Prospective Randomized Clinical Trial. Obes Surg. 2016 Nov;26(11):2616-2621. doi: 10.1007/s11695-016-2142-z. PMID 27007272
- [Background] Yong L, Guang B. Intraperitoneal ropivacaine instillation versus no intraperitoneal ropivacaine instillation for laparoscopic cholecystectomy: A systematic review and meta-analysis. Int J Surg. 2017 Aug;44:229-243. doi: 10.1016/j.ijsu.2017.06.043. Epub 2017 Jun 30. PMID 28669869

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT07400146/Prot_SAP_000.pdf
  • Informed Consent Form (2026-01-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT07400146/ICF_001.pdf